CLINICAL TRIAL: NCT02538328
Title: Comparison of Harmonic Scalpel and Ligasure Devices in Laparoscopic Morbid Obesity Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Serdar Kırmızı, General Surgeon in Gastrointestinal Surgery, Inonu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 2014/105
Record Dates: First submitted 2015-08-10; First posted 2015-09-02 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-08

CONDITIONS: Morbid Obesity
Keywords: laparoscopy; obesity; harmonic scalpel; ligasure
MeSH Terms: conditions — Obesity, Morbid; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- harmonic scapel (Active Comparator): Obesity surgery cases where hamonic scalpel is used for the comparison of different surgical devices
  Interventions: Device: Harmonic scapel; Device: Ligasure
- Ligasure sealing device (Placebo Comparator): Ligasure used in obesity surgery for the comparison of different surgical devices Randomly chosen cases where ligasure is used instead of hamonic scalpel in surgical procedures comparison of multiple dissectors
  Interventions: Device: Harmonic scapel; Device: Ligasure

INTERVENTIONS:
Device: Harmonic scapel — different surgical devices used in the obesity surgery
  Other Names: ultrasonic dissector
Device: Ligasure — Bipolar vessel sealing system used in obesity surgery
  Other Names: Bipolar Vessel sealing device

SUMMARY:
Comparison of harmonic scalpel and ligasure devices in laparoscopic morbid obesity surgery especially in gastric bypass surgery patients.

DETAILED DESCRIPTION:
The investigators' department performs 150 gastric bypass surgeries annually. Surgeons use both harmonic scalpel and ligasure sealing device in cases. Aim is to compare both of these devices over coming each other. Benefits ease of these devices are compared.

ELIGIBILITY:
Inclusion Criteria:

* obesity
* BMI over 40 kg/m^2

Exclusion Criteria:

* Normal BMI cases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2014-07; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Safety and efficacy of sealing | 1 year
  Aim to compare the fogging and the time spend performing the gastric resection to form the gastric pouch.

SECONDARY OUTCOMES:
Bleeding | During the operation
  Amount of blood loss in the operation

CONTACTS AND LOCATIONS:
Overall Officials: cüneyt kayaalp, prof, Principal Investigator — GENERAL SURGERY CHİEF OF GASTROİNTESTİNAL SURGERY